CLINICAL TRIAL: NCT05875844
Title: Effectiveness of Wrist Splint and Occupational Therapy to Improve Pain, Mobility and Functional Status in Patients With Wrist Drop
Brief Title: Wrist Splint and Occupational Therapy to Improve Pain, Mobility and Functional Status in Patients With Wrist Drop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/545
Record Dates: First submitted 2023-03-18; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Wrist-Drop
MeSH Terms: conditions — Radial Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wrist Splint (Other)
  Interventions: Diagnostic Test: Wrist Splint
- Occupational Therapy (Experimental)
  Interventions: Diagnostic Test: Occupational Therapy

INTERVENTIONS:
Diagnostic Test: Wrist Splint — Wrist Splint to Improve Pain, Mobility and Functional Status in Patients With Wrist Drop
  Arms: Wrist Splint
Diagnostic Test: Occupational Therapy — Occupational Therapy to Improve Pain, Mobility and Functional Status in Patients With Wrist Drop
  Arms: Occupational Therapy

SUMMARY:
To determine effectiveness of wrist splint and occupational therapy to improve pain, mobility and functional status in patients with wrist drop.

ELIGIBILITY:
Inclusion Criteria:

* • People with wrist drop

  * People between 20 to 40 years will be included (male and female)
  * Post-operative patients (nerve grafting and plastic surgery)
  * Patients with findings of nerve compression will be included

Exclusion Criteria:

* • People with nerve injuries other than radial nerve such as ulnar or median nerve

  * People suffering with other neurological disorders.
  * People who are not able to follow instructions
  * Any traumatic history
  * Diabetic patients, thyroid issues, pregnant females

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
DASH scale (0-100) | 6 Months
  DASH questionnaire for function on the scale of (0-100) worst zero- hundred normal
VAS on the scale (1-10) | 6 Months
  VAS for pain for pain (0-10) 0 for normal, 10 for worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No